CLINICAL TRIAL: NCT05557370
Title: Prospective Analysis of Immunogenicity of the Nonavalent Human Papillomavirus Vaccination (GARDASIL 9) in Patients Post Solid Organ Transplant
Brief Title: Immunogenicity of HPV Vaccine in Transplant Recipients.
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Denise Uyar, Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HPV MK-MISP 61451
Record Dates: First submitted 2022-09-14; First posted 2022-09-28 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Diseases; Kidney Transplant
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Papillomavirus Vaccines; Human Papillomavirus Recombinant Vaccine nonavalent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Interventional (Experimental): Patient between the age of 18 and 45 years with at least 6 months post-solid-organ transplant who has not received GARDASIL 9.
  Interventions: Biological: Human Papilloma Virus vaccine (GARDASIL 9)

INTERVENTIONS:
Biological: Human Papilloma Virus vaccine (GARDASIL 9) — Patients will be scheduled to receive 3-dose 9vHPV vaccination (vaccination at enrollment [time 0], 2 months [+ 6 weeks], and 6 months [+ 6 weeks] per standard guidelines).

SUMMARY:
To measure levels of HPV antibodies in post-solid-organ transplant recipients who have gotten the HPV9 vaccine.

DETAILED DESCRIPTION:
This is a prospective open-label nonrandomized single-center cohort study aimed to analyze the immunogenicity of nanovalent human papillomavirus vaccination (GARDASIL 9) in post-solid-organ transplant patients.

The study duration is anticipated to be 36 months. The expected duration of subject participation is 24 months. Immunocompromised populations are at greater risk of HPV infection. Quadrivalent HPV vaccination has been performed and lower titers of antibodies have been compared to published date in non-immunocompromised population (controls). The HPV9 vaccination titers have not been measured in the immunocompromised population to date.

We plan to enroll 30 adult solid-organ transplant recipients ages 18-45 years >6 months from transplant receiving treatment at clinics at F&MCW Main Campus.

Patients will be scheduled to receive 3-dose 9vHPV vaccination (vaccination at enrollment [time 0], 2 months [+ 6 weeks], and 6 months [+ 6 weeks] per standard guidelines).

Serial serum samples will be obtained for geometric mean titers (GMT) prior to vaccination, at 7 months (+ 6 weeks), 12 months (+ 6 weeks), and 24 months (+ 6 weeks) after completion of the vaccination series. If a patient is subsequently scheduled to undergo a transplant, we will obtain the GMT prior to the transplant.

Subjects will be asked to consent to optional banking of whole-blood for future research and translational studies. Blood will be stored in the Obstetrics & Gynecology Specimen and Data Bank (PRO 11631) at Medical College of Wisconsin.

If subjects chose to participate in the optional banking of their blood, approximately 5 mls of additional blood will be drawn prior to vaccination and at the time of the 7, 12, and 24- month GMT blood draws.

Anti-HPV antibody responses will be measured using a proprietary MERCK Competitive Luminex Immunoassay (cLIA) which will be performed by Merck and expressed as geometric mean titers (GMT).

ELIGIBILITY:
Inclusion Criteria:

1. Patient between the age of 18 and 45 years
2. Patient is at least 6 months post-solid-organ transplant and has not received GARDASIL 9.
3. Patient who can participate in their health care and sign informed consent.
4. Patient may have had bivalent or quadrivalent HPV vaccination previously.
5. Living or deceased donor transplant patient is eligible.

   Exclusion Criteria:
6. Contraindication: Hypersensitivity, including severe allergic reactions to yeast (a vaccine component), or after a previous dose of GARDASIL 9 or GARDASIL.
7. Patient had completed vaccination series with a nonavalent HPV vaccine (e.g., GARDASIL 9) in the past
8. Patient with a diagnosis of HIV.
9. Patient that endorses being currently pregnant.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 7 months, 12 months and 24 months
  The primary outcome is to measure immunogenicity using the Merck proprietary Competitive Luminex Immunoassay (cLIA) and geometric mean titers (GMTs) over specified time intervals (7 months, 12 months and 24 months from vaccination) in patients to each of the nine human papillomavirus types contained in the nanovalent human papillomavirus vaccine (HPV9) vaccination and compare these antibody levels to published control data for non-immunocompromised individuals. this has been completed previously for the quadrivalent HPV vaccination series but no data exists for the HPV9 vaccination in this population.
  We will also compare GMTs in our study patients and over time to determine if there is a difference between timing of vaccine administration.

SECONDARY OUTCOMES:
Secondary Outcome | 7 months, 12 months and 24 months
  Immunogenicity using the Merck proprietary Competitive Luminex Immunoassay (cLIA) and geometric mean titers (GMTs) over specified time intervals (7 months, 12 months and 24 months from vaccination) in a patient cohort prior to kidney. We will assess the change in GMT over time.
  The utilization of regression analysis to determine the effect of variables on antibody response (GMTs) such as age, gender, race, renal function and type of immunosuppression, and donor type.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Uyar, MD, Principal Investigator — Medical College of Wisconsin/ Froedtert Hospital
Locations (1):
- Froedtert Lutheran Memorial Hospital, Milwaukee, Wisconsin, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/70/NCT05557370/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/70/NCT05557370/ICF_001.pdf